CLINICAL TRIAL: NCT01014182
Title: Early Invasive Strategy After Fibrinolysis vs Standard Management in STEMI Patients: Results From an Individual Patient Data Meta-analysis (OTTER Meta-analysis) OTTER: Optimal Timing for Post-Thrombolysis Elective Revascularization
Brief Title: Early Percutaneous Coronary Intervention (PCI) After Fibrinolysis Versus Standard Therapy in ST Segment Elevation Myocardial Infarction (STEMI) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Prof.Carlo Di Mario, Royal Brompton & Harefield NHS Foundation Trust
Other Study IDs: OTTER220179
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2009-11-16 (Estimated); Status verified 2009-11

CONDITIONS: Myocardial Infarction
Keywords: Early PCI; Myocardial Infarction; Thrombolysis; Optimal revascularization therapy in STEMI patients
MeSH Terms: conditions — Myocardial Infarction

GROUPS / COHORTS (2):
- Early PCI: Routine invasive strategy with early PCI performed in STEMI patients within 24 hours from successful fibrinolysis
- Standard Therapy: Standard therapy in STEMI patients with fibrinolysis and/or conventional ischaemic-guided therapy.

SUMMARY:
Several recent trials (1,2) suggest that all STEMI patients receiving fibrinolysis in non-PCI centres should be routinely transferred for elective early PCI within 24 hours from hospitalization, with no additive risk of major bleeding complications or other severe adverse events compared standard therapy. These results in favour of a routine invasive strategy in STEMI patients suggest a potential change to the current approach of awaiting the response to treatment in patients receiving fibrinolysis, and draw the attention to the potential need for an appropriate network organization with adequate first hospitalization treatment (spoke) and prompt transfer to centres with 24/7 PCI capabilities (hub). The recent ESC (3) and ACC (4) guidelines on STEMI are consistent with the early ESC PCI Guidelines, recommending that angioplasty after fibrinolysis should be performed within a time-window ranging between 3 and 24 hours after successful lytic administration (level evidence IIA). The reason for the weighting of the recommendation is due to the heterogeneity of trial results with different planned-revascularization strategies, variable primary end-points definitions, and small individual trial sample sizes. Therefore, a consistent analysis of single patient dataset from all published randomized trials would be of value to better define the magnitude and duration of clinical benefit of the routine invasive strategy after lytic treatment as well as the potential optimal timing of such a strategy.

The main aim of the OTTER meta-analysis is to define the benefits of immediate PCI after fibrinolysis for STEMI patients. Moreover, the OTTER meta-analysis will investigate the optimal timing of post-fibrinolysis elective revascularization.

DETAILED DESCRIPTION:
All published randomized controlled trials that compared a routine invasive strategy with early PCI and a standard therapy in STEMI patients after fibrinolysis will be included in this analysis.

We will exclude all non-randomized trials, randomized studies if the individual patient data will not be available for analysis, randomized studies in which angioplasty was mainly performed without stenting (<80% stenting population) and in which the type of lytic therapy was different from modern fibrin-specific agents. Two investigators independently will evaluate studies for possible inclusion. The quality of searched trials will be evaluated based on the 5-point scale outlined by Jadad et al (5), with criteria for randomization with proper concealment of the allocation sequence, blinding of the patient and investigators to treatment allocation with description of the blinding method, and completeness of follow-up.

Recruitment:

An electronic database will be compiled consisting of data from each single patient of all enrolled trials, according to the guidelines for the performance of individual patient meta-analysis.(6-7-8). The database will include demographic data and baseline characteristics. Attention will be paid to clinical complications during transfer for early PCI and to the precise calculation of the following times-window: from symptoms onset to lytic therapy, from lytic therapy to early or rescue PCI, from randomization to all adverse events as defined below. Data will be checked for completeness and for consistency with published reports. Two investigators independently will extract all data, with disagreements resolved in consultation with a third investigator.

End-points

The following end-points will be investigated:

Primary End Point: Combined death/reinfarction at 30 days.

Secondary end-points:

* Death, reinfarction, recurrent ischemia and urgent revascularization at 30 days.
* Combined death/reinfarction/recurrent ischemia/urgent revascularization and new presentation CHF and shock at 30 days.
* Major bleeding and hemorrhagic stroke at 30 days.
* Combined death/reinfarction and combined revascularization/recurrent ischemia at 6-12 months.

Secondary analysis will also investigate the influence of the timing of post-thrombolysis early revascularization on the above considered events.

Investigators: The study is coordinated by Prof. C. Di Mario. An executive committee composed of the Principle Investigators of the enrolled trials will overview the quality of data collected (OTTER Investigators). No publication will be sent without written consent of all the PIs of the individual trials. Statistical analysis will be performed at the Royal Brompton Hospital (London) and the Canadian Heart Research Centre (Toronto, Ontario, Canada).

References:

1. Cantor WJ, Fitchett D, Borgundvaag B, Ducas J, et al. TRANSFER-AMI Trial Investigators. Routine early angioplasty after fibrinolysis for acute myocardial infarction. N Engl J Med. 2009 Jun 25;360(26):2705-18.
2. Di Mario C, Dudek D, Piscione F, et al. Immediate angioplasty versus standard therapy with rescue angioplasty after thrombolysis in the Combined Abciximab REteplase Stent Study in Acute Myocardial Infarction (CARESS-in-AMI): an open, prospective, randomized, multicentre trial. Lancet 2008; 371:559-568.
3. Van de Werf F, Bax J, Betriu A, et al. Management of acute myocardial infarction in patients presenting with persistent ST-segment elevation: the Task Force on the Management of ST-Segment Elevation Acute Myocardial Infarction of the European Society of Cardiology. Eur Heart J 2008; 29:2909-2945.
4. Antman EM, Hand M, Armstrong PW, et al. 2007 focused update of the ACC/AHA 2004 guidelines for the management of patients with ST-elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol 2008; 51:210-247.
5. Jadad AR, Moore RA, Carroll D, et al. Assessing the quality of reports of randomized clinical trials: is blinding necessary? Control Clin Trials. 1996 Feb;17(1):1-12.
6. Simmonds MC, Higgins JP, Stewart LA, et al. Meta-analysis of individual patient data from randomized trials: a review of methods used in practice. Clin Trials. 2005;2(3):209-17.
7. Clarke MJ, Stewart LA. Meta-analyses using individual patient data. J Eval Clin Pract. 1997 Aug;3 (3):207-12. Review. PubMed PMID: 9406108
8. Stewart LA, Clarke MJ. Practical methodology of meta-analyses (overviews) using updated individual patient data. Cochrane Working Group. Stat Med. 1995 Oct 15;14(19):2057-79.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients enrolled within 12 hours from onset of symptoms
* Controlled randomized trials comparing a routine invasive strategy with standard therapy in STEMI patients
* Modern fibrin-specific therapy in both groups
* Stenting PCI > 80% of invasive procedures
* English language

Exclusion Criteria:

* Cardiogenic shock at presentation
* Need for concomitant
* Major surgery
* Severe chronic renal or hepatic impairment
* Myocardial infarction within the previous 2 weeks
* Contraindications to thrombolytic therapy, abciximab, aspirin, or clopidogrel
* Non randomized trials
* Single patient data not available
* Non fibrin-specific lytic therapy
* Stenting PCI < 80% of invasive procedures
* Not English language

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: STEMI patients.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2009-11; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Combined death/reinfarction | 30 days

SECONDARY OUTCOMES:
Death, reinfarction, recurrent ischemia and urgent revascularization | 30 days
Combined death/reinfarction/recurrent ischemia/urgent revascularization and new presentation CHF and shock | 30 days.
Major bleeding and hemorrhagic stroke | 30 days
Combined death/reinfarction and combined revascularization/recurrent ischemia | 6-12 months
Influence of Optimal Timing of Post-Thrombolysis early revascularization on primary and secondary clinical end-points | 0-24 hours from thrombolysis

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

REFERENCES:
- [Derived] Abdel-Qadir H, Yan AT, Tan M, Borgia F, Piscione F, Di Mario C, Halvorsen S, Cantor WJ, Westerhout CM, Scheller B, Le May MR, Fernandez-Aviles F, Sanchez PL, Lee DS, Goodman SG. Consistency of benefit from an early invasive strategy after fibrinolysis: a patient-level meta-analysis. Heart. 2015 Oct;101(19):1554-61. doi: 10.1136/heartjnl-2015-307815. Epub 2015 Jul 14. PMID 26175478
- [Derived] Madan M, Halvorsen S, Di Mario C, Tan M, Westerhout CM, Cantor WJ, Le May MR, Borgia F, Piscione F, Scheller B, Armstrong PW, Fernandez-Aviles F, Sanchez PL, Graham JJ, Yan AT, Goodman SG. Relationship between time to invasive assessment and clinical outcomes of patients undergoing an early invasive strategy after fibrinolysis for ST-segment elevation myocardial infarction: a patient-level analysis of the randomized early routine invasive clinical trials. JACC Cardiovasc Interv. 2015 Jan;8(1 Pt B):166-174. doi: 10.1016/j.jcin.2014.09.005. Epub 2014 Oct 31. PMID 25616922